CLINICAL TRIAL: NCT04824313
Title: Vascular Abnormalities Detected With Chest CT in COVID-19: Spectrum, Association With Other Lesions, and Correlation With Clinical Severity
Brief Title: Vascular Abnormalities Detected With Chest CT in COVID-19
Acronym: COVID-CAVA
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Salah D. Qanadli (Other)
Collaborators: University of Geneva, Switzerland (Other); University of Bern (Other); University of Basel (Other); University of Zurich (Other)
Responsible Party: Sponsor-Investigator, Salah D. Qanadli, Prof. MD, PhD, University of Lausanne
Organization: University of Lausanne (Other)
Other Study IDs: 2020-1469
Record Dates: First submitted 2021-02-18; First posted 2021-04-01 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Covid19; Pneumonia, Viral; Pulmonary Embolism
Keywords: COVID-19; Computed tomography; Vascular abnormalities; Lung infection; Thromboembolism
MeSH Terms: conditions — COVID-19; Pneumonia, Viral; Pulmonary Embolism; Thromboembolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 6 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COVID-CAVA PE: Patients with RT-PCR proven COVID-19 disease and CTA proven pulmonary embolism
  Interventions: Diagnostic Test: Chest CTA
- COVID-CAVA non-PE: Patients with RT-PCR proven COVID-19 disease and no evidence of pulmonary embolism on CT
  Interventions: Diagnostic Test: Chest CT; Diagnostic Test: Chest CTA

INTERVENTIONS:
Diagnostic Test: Chest CT — Chest CT without intravenous contrast material
  Groups: COVID-CAVA non-PE
Diagnostic Test: Chest CTA — Chest CT with intravenous contrast material

SUMMARY:
Chest computed tomography of patients having coronavirus disease (COVID-19) will be analyzed with regards to vascular abnormalities (pulmonary embolism and vascular thickening), and their association with lung inflammation. The prevalence, severity, distribution, and prognostic value of chest CT findings will be assessed. Patients with vascular abnormalities will be compared to patients without, which is supposed to provide insights into the prognostic role of such abnormalities, and the potential impact on treatment strategy.

DETAILED DESCRIPTION:
Since the SARS-CoV-2 outbreak, computed tomography (CT) imaging has almost immediately established itself as the primary non-invasive diagnostic tool for diagnosis, monitoring of COVID-19 pneumonia, and complications thereof.

While most of the currently available literature relies on non-contrast CT, the need to assess vascular abnormalities is being recognized as an increasingly important factor, both to help distinguish COVID-19 pneumonia from other viral infections, and to exclude pulmonary embolism (PE). Acute PE is believed to be a significant contributory factor in patients with adverse outcomes.

Relating to vascular changes other than PE, additional knowledge is required and not yet available to confirm and better understand early observations. In particular, a radiological sign referred to as "vascular thickening", "vascular enlargement", or "vascular congestion" that is thought to be a specific marker of COVID-19 pneumonia, calls for a thorough assessment. Quantitative analysis of this sign and correlation to clinical presentation is highly desirable.

The investigators will conduct a multicentric observational study in the form of a registry. For this purpose, each participating center needs to screen hundreds of COVID-19 patients to select those who meet the inclusion criteria and do not have any exclusion criteria. Then, clinical, laboratory and imaging data of eligible patients will be retrieved. The research will focus on the imaging manifestations of COVID-19 pneumonia and their relationship to vascular abnormalities within the lung; the potential association between such vascular abnormalities and COVID-19 clinical severity will be assessed.

To achieve adequate statistical power, the study needs to be multicentric, involving 7 Swiss institutions; CHUV Lausanne, USZ Zurich, USB Basel, Inselspital Bern, Division Stadt- und Landspitäler Inselgruppe, HUG Genève, HRC Rennaz. The following investigators are involved in this extensive nationwide effort:

* CHUV: Dr DC Rotzinger; Prof SD Qanadli; Prof PY Bochud; Prof L Alberio; Dr JL Pagani
* USZ: Prof H Alkadhi
* USB: Prof J Bremerich; Dr A Sauter
* Inselspital: Prof T Heverhagen; Prof L Ebner
* Division Stadt- und Landspitäler Inselgruppe: Prof A Christe
* HUG: Prof A Poletti
* HRC: Prof O Ratib

Intrahospital medical records, laboratory tests results, and data from chest CT performed in the participating centers between March 1st and July 31st, 2020 will be used to:

* assess the frequency of non-PE related vascular abnormalities on chest CT (vascular thickening), and their association with parenchymal opacities
* evaluate the rate of acute PE among the patients undergoing contrast-enhanced chest CT
* quantify the clot burden in terms of proximal or distal obstruction and quantitative CT obstruction index (CTOI) in patients with CT-proven PE
* evaluate the consequence of PE on pulmonary perfusion (distinguishing perfused vs. non-perfused pulmonary opacities) and cardiac morphology (right ventricle dilatation, reduced left atrial size)
* evaluate the correlation between pulmonary perfusion impairment and clinical severity

Using clinical, laboratory and CT imaging-derived variables, the investigators will perform outcome modelling to derive an integrative score to predict outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted for COVID-19 (with positive rt-PCR for SARS-CoV-2) who had a contrast-enhanced chest CT within the specified timeframe.

Exclusion Criteria:

* Age <18 years Patients with another pre-existing infectious process Documented refusal of the reuse of medical data

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients with positive rt-PCR for SARS-CoV-2 and chest CT (with or without intravenous contrast material injection) within the specified time frame.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2021-03-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of acute pulmonary embolism | March 1st, 2020 to July 31st, 2020
  Incidence of acute pulmonary embolism (PE).
Distribution of acute pulmonary embolism | March 1st, 2020 to July 31st, 2020
  Description of the anatomical distribution (lobar and segmental level)
Pulmonary embolism clot burden | March 1st, 2020 to July 31st, 2020
  Description of the clot burden of acute pulmonary embolism (PE) using the CT obstruction index
Association of pulmonary embolism with ground glass opacity | March 1st, 2020 to July 31st, 2020
  Rate of PE in segments with vs. without COVID-19 ground glass opacity

SECONDARY OUTCOMES:
Clinical outcome | March 1st, 2020 to July 31st, 2020
  Outcome will be registered in a categorical variable as outpatient, inpatient without intubation, inpatient with intubation, death
D-dimers | March 1st, 2020 to July 31st, 2020
  D-dimer serum sampling (ng/mL), continuous variable
PO2 | March 1st, 2020 to July 31st, 2020
  Arterial blood oxygen partial pressure (PO2, mmHg), continuous variable
SaO2 | March 1st, 2020 to July 31st, 2020
  Venous blood oxygen saturation (SaO2, in %), continuous variable
CRP | March 1st, 2020 to July 31st, 2020
  C-reactive protein serum sampling (mg/L), continuous variable
Thrombocytes | March 1st, 2020 to July 31st, 2020
  Blood thrombocyte count (number per liter), continuous variable
ICU admission | March 1st, 2020 to July 31st, 2020
  Rate of patients admitted in the intensive care unit (ICU)
Alveolar opacity | March 1st, 2020 to July 31st, 2020
  Rate of lung segments with alveolar opacity
Vascular congestion | March 1st, 2020 to July 31st, 2020
  Rate of lung segments with vascular congestion
Vascular volume | March 1st, 2020 to July 31st, 2020
  Vascular volume measured at the segmental level (in mL), continuous variable
Vein-to-artery ratio | March 1st, 2020 to July 31st, 2020
  The vein-to-artery ratio will be calculated at the segmental level (venous diameter [mm] / arterial diamter [mm]), continuous variable

CONTACTS AND LOCATIONS:
Locations (1):
- CHUV, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Qanadli SD, Beigelman-Aubry C, Rotzinger DC. Vascular Changes Detected With Thoracic CT in Coronavirus Disease (COVID-19) Might Be Significant Determinants for Accurate Diagnosis and Optimal Patient Management. AJR Am J Roentgenol. 2020 Jul;215(1):W15. doi: 10.2214/AJR.20.23185. Epub 2020 Apr 7. No abstract available. PMID 32255684
- [Derived] Nevesny F, Rotzinger DC, Sauter AW, Loebelenz LI, Schmuelling L, Alkadhi H, Ebner L, Christe A, Platon A, Poletti PA, Qanadli SD. Acute Pulmonary Embolism in COVID-19: A Potential Connection between Venous Congestion and Thrombus Distribution. Biomedicines. 2022 Jun 2;10(6):1300. doi: 10.3390/biomedicines10061300. PMID 35740322